CLINICAL TRIAL: NCT02188004
Title: The Epidemiologic Study of Human Papillomavirus Infection and Related Diseases In Male and Female Aged Over 18 Years In China
Brief Title: The Epidemiologic Study of Human Papillomavirus Infection and Related Diseases
Status: Completed | Type: Observational
Sponsor: Jun Zhang (Other)
Collaborators: Liuzhou center of disease prevention and control (Unknown)
Responsible Party: Sponsor-Investigator, Jun Zhang, professor, Xiamen University
Organization: Xiamen University (Other)
Other Study IDs: HPV-EPI-001
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Human Papillomavirus Infection; Genital Warts
Keywords: HPV; genital warts
MeSH Terms: conditions — Papillomavirus Infections; Condylomata Acuminata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Male:Two swabs were used to collect exfoliated skin cells from the coronal sulcus /glans/shaft and anal
  Female:Three swabs were used to collect exfoliated skin cells from the vagina，vulva and anal
Oversight: Data Monitoring Committee: No

SUMMARY:
primary purpose:Evaluate the prevalence and incidence of HPV infection and related diseases in subjects.

Secondary purpose:Analyze risk factors of HPV infection and related diseases.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 55 years;
* residents of the study site;
* at least one sex partner;
* Be able to understand and comply with the request of the protocol.

Exclusion Criteria:

* pregnant;
* has received HPV vaccines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 5000 healthy volunteers will be recruited from the residents of Liuzhou through advertisment.
Sampling Method: Non-Probability Sample
Enrollment: 4691 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
prevalence and incidence of HPV infection | 1 year
  Evaluate the prevalence and incidence of HPV infection and related diseases in subjects

SECONDARY OUTCOMES:
risk factors of HPV infection and related diseases | 1 year
  Analyze risk factors of HPV infection and related diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Study Chair — Xiamen University; Ming-Qiang Li, Principal Investigator — Liuzhou center of disease prevention and control
Locations (1):
- Liuzhou Center of disease prevention and control, Liuchow, Guangxi, China

REFERENCES:
- [Derived] Wei F, Guo M, Huang S, Li M, Cui X, Su Y, Wu X, Ma X, Zheng Y, Huang Y, Wang L, Pan L, Wu T, Zhang J, Xia N. Sex Differences in the Incidence and Clearance of Anogenital Human Papillomavirus Infection in Liuzhou, China: An Observational Cohort Study. Clin Infect Dis. 2020 Jan 1;70(1):82-89. doi: 10.1093/cid/ciz168. PMID 30852604